CLINICAL TRIAL: NCT04580524
Title: Poly-4-hydroxybutyrate Mesh Versus Current Care of Complex Open Ventral Hernias: A Multi-Center Randomized Controlled Trial
Brief Title: Phasix Mesh Use in Complex Open Ventral Hernias Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not able to secure funding
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Julie Holihan, Assistant Professor of Surgery-Clinical, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-20-0655
Record Dates: First submitted 2020-10-02; First posted 2020-10-08 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phasix Mesh (Active Comparator): Phasix mesh will be used in the repair of the hernia
  Interventions: Procedure: Repair of ventral hernia using biologic mesh
- Current Care (Active Comparator): The hernia will be repaired with either synthetic mesh or suture repair, as determined by the operating surgeon.
  Interventions: Procedure: Repair of ventral hernia using suture repair or synthetic mesh

INTERVENTIONS:
Procedure: Repair of ventral hernia using biologic mesh — Ventral hernia will be repaired using biologic mesh
  Arms: Phasix Mesh
Procedure: Repair of ventral hernia using suture repair or synthetic mesh — Ventral hernia will be repaired using the current treatment methods
  Arms: Current Care

SUMMARY:
The purpose of this study is to compare clinical and patient centered outcomes of biosynthetic poly-4-hydroybutyrate meshes versus current care (synthetic polypropylene mesh or suture) for complex ventral hernia repair. The primary outcome for this study will be patients who are major complication free at 2 years postoperative. This will be a composite of hernia recurrence, reoperation, chronic wound complication, or death. Secondary outcomes include: surgical site occurences such as surgical site infection, seroma, hematoma and skin dehiscence within 90 days postoperative, emergency room visits withing 90 days postoperative, days in hospital up to 90 days postoperative, abdominal pain, and change in patient centered outcomes measured through the modified activities assessment scale (mAAS).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years or older) with a complex ventral hernia scheduled for repair

Exclusion Criteria:

* Patients likely to die within 3 years (cirrhosis, terminal cancer, surgeon judgement)
* Unlikely to follow-up (live out of state, unable to be reached by phone or email)
* Non-English and non-Spanish speakers
* Pregnant or breast-feeding patients
* Allergies/hypersensitivities to tetracycline hydrochloride and kanamycin sulfate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Major complication free | 2 years post-operative
  A composite of hernia recurrence, reoperation, chronic wound complication, or death

SECONDARY OUTCOMES:
Surgical site occurrences | 90 days post-operative
  Surgical site infection, seroma, hematoma, and skin dehiscence
Clavien-Dindo complication grade | 90 days post-operative
  Clavien-Dindo complication grade
Hospital duration | 90 days post-operative
  Days in hospital composed of post-operative length of stay and readmissions
Emergency room visits | 90 days post-operative
  Number of times ER was visited
Cost Analysis | 2 years
  Analysis of costs as performed from the healthcare perspective
Post-operative abdominal pain | Day of consent and post-operatively at 1 month, 1 year and 2 years
  Measured by the visual analogue scale (VAS)
Patient centered outcomes | Day of consent and post-operatively at 1 month, 1 year and 2 years
  Abdominal wall health status (AW-HS) measured through the modified activities assessment scale (mAAS)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Holihan, MD, Principal Investigator — UTHealth
Locations (2):
- United States (2):
  - Lyndon B. Johnson General Hospital, Houston, Texas
  - Memorial Hermann Hospital-Texas Medical Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No